CLINICAL TRIAL: NCT04648215
Title: The Effect of Lavender Aromatherapy on Sleep in Hospitalized Adult Patients
Brief Title: Lavender Aromatherapy for Sleep in Hospitalized Adult Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unavailable subjects
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-0423
Record Dates: First submitted 2020-11-03; First posted 2020-12-01 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Sleep; Hospitalization
Keywords: lavender aromatherapy, sleep
MeSH Terms: interventions — lavender oil

STUDY DESIGN:
Intervention Model Description: Randomized three group design : lavender aromatherapy (intervention); grapeseed oil aromatherapy (placebo) ; standard of care for night time (control)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- lavender oil (Experimental): lavender oil as aromatherapy two drops dispensed on a 2x2 gauze and pinned to subject's gown
  Interventions: Other: lavender oil
- grapeseed oil (Placebo Comparator): grapeseed oil as aromatherapy two drops dispensed on a 2x2 gauze and pinned to subject's gown
  Interventions: Other: Grapeseed Oil
- Standard of Care (No Intervention): Routine nursing care at bedtime (HS)

INTERVENTIONS:
Other: lavender oil — aromatherapy--two drops applied to a 2x2 gauze and pinned to subject's gown
  Arms: lavender oil
Other: Grapeseed Oil — aromatherapy--two drops applied to a 2 X 2 gauze and pinned to subject's gown
  Arms: grapeseed oil

SUMMARY:
This feasibility study's aim is to determine the effectiveness of lavender oil aromatherapy on quality and duration of sleep in hospitalized adult patients

DETAILED DESCRIPTION:
Hospitalized patients on a medical unit will be randomly assigned to one of three groups of 36 patients: Intervention (Lavender oil), Placebo Intervention (Grapeseed Oil), or Control (Standard of Care). Following a determination of meeting inclusion criteria on admission and completing informed consent, subjects will be randomized to one of three groups on admission. This is a 4 day study with pre- intervention (baseline) sleep data on quality and duration of sleep using the Verrans & Halpern- Snyder Sleep Scale collected on Day 2, following admission day.

For the intervention, indirect aromatherapy, a 2x2 gauze with 2 drops of either oil (lavender or grapeseed is pinned it to the subjects' nightgown (right scapula area) for two sequential nights (Time 1 and Time 2) (Day 2 and 3) and removed in the morning after 10 hours . Sleep Quality and Duration are then measured in the morning, Time 1 and Time 2, (Day 3 and Day 4) by the Verran & Snyder-Halpern Sleep Scale analogue. The control group receives standard of care in the evenings and the same data as the intervention groups are collected for sleep quality and duration, pre-intervention and Time 1 and Time 2 ..

The differences in the scores for sleep quality and duration will be compared from pre-intervention to Time 1 and Time 2 for each group .

ELIGIBILITY:
Inclusion Criteria

* Ability to speak, read and understand English.
* Ability to use an electronic "pad" following instruction and assistance for data collection

Exclusion Criteria:

* Cognitive impairment .Allergy to lavender or grapeseed oil
* .Any condition that has been reported to affect the sense of smell
* Newly prescribed sleep medications (last two weeks prior to admission) or those causing sleepiness
* Pregnancy
* Currently using lavender therapy (aroma, massage, etc.).
* A smoker of any kind (tobacco, electronic cigarettes) .
* History of migraine headaches.
* Asthma, Bronchitis, or any airway disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in sleep duration from Baseline to Day 3 and day 4 | Baseline, Day 3, Day 4
  Measured by an increase in the mean scores Verans and Snyder-Halpern Sleep Scale (0-100) by 10 or greater
Change in sleep quality from Baseline to Day 3 and Day 4 | Baseline Day 3, Day 4
  Measured by an increase in mean scores on the the Verans and Snyder-Halpern Sleep Scale of 10 or greater

CONTACTS AND LOCATIONS:
Overall Officials: Jane H. White, PhD, Principal Investigator — Northwell Health, Nurse Scientist IFN
Locations (2):
- United States (2):
  - Northwell Health , South Shore University Hospital, Bay Shore, New York
  - South Shore University Hosp, Bay Shore, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stepanski EJ, Wyatt JK. Use of sleep hygiene in the treatment of insomnia. Sleep Med Rev. 2003 Jun;7(3):215-25. doi: 10.1053/smrv.2001.0246. PMID 12927121
- [Background] Tamrat R, Huynh-Le MP, Goyal M. Non-pharmacologic interventions to improve the sleep of hospitalized patients: a systematic review. J Gen Intern Med. 2014 May;29(5):788-95. doi: 10.1007/s11606-013-2640-9. Epub 2013 Oct 10. PMID 24113807
- [Background] Tranmer JE, Minard J, Fox LA, Rebelo L. The sleep experience of medical and surgical patients. Clin Nurs Res. 2003 May;12(2):159-73. doi: 10.1177/1054773803012002004. PMID 12741668
- [Result] Cho EH, Lee MY, Hur MH. The Effects of Aromatherapy on Intensive Care Unit Patients' Stress and Sleep Quality: A Nonrandomised Controlled Trial. Evid Based Complement Alternat Med. 2017;2017:2856592. doi: 10.1155/2017/2856592. Epub 2017 Dec 11. PMID 29375641
- [Result] Dobing S, Frolova N, McAlister F, Ringrose J. Sleep Quality and Factors Influencing Self-Reported Sleep Duration and Quality in the General Internal Medicine Inpatient Population. PLoS One. 2016 Jun 9;11(6):e0156735. doi: 10.1371/journal.pone.0156735. eCollection 2016. PMID 27280292
- [Result] Park MJ, Yoo JH, Cho BW, Kim KT, Jeong WC, Ha M. Noise in hospital rooms and sleep disturbance in hospitalized medical patients. Environ Health Toxicol. 2014 Aug 18;29:e2014006. doi: 10.5620/eht.2014.29.e2014006. eCollection 2014. PMID 25163680